CLINICAL TRIAL: NCT04584099
Title: Histological Study to Assess Safety and Efficacy of the TempSure Firm for Non-invasive Lipolysis
Brief Title: Multi-Center Traditional Feasibility Study of Radiofrequency Device
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study stopped due to a business decision.
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CYN20-FIRM-HISTO
Record Dates: First submitted 2020-09-24; First posted 2020-10-12 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Body Fat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Biopsy Removed Post Tx (Experimental): All subjects had one radiofrequency treatment before scheduled biopsy or abdominoplasty on tissue to be removed during abdominoplasty immediately post treatment, 10 days post treatment, 20 days post treatment, and/or 30 days post treatment.
  Interventions: Device: Radiofrequency device treatment

INTERVENTIONS:
Device: Radiofrequency device treatment — TempSure firm

SUMMARY:
This is a prospective, controlled, multi-center study. Patients will be enrolled and treated with a radiofrequency device in this study if they have unwanted fat in the abdominal area.

DETAILED DESCRIPTION:
Subjects are to be enrolled in this clinical study if they are 18 - 55 years old and are willing to have biopsies taken from a control site and the treatment area. Subjects may be enrolled if they have been previously scheduled or willing to have an abdominoplasty procedure after their participation in the study. A maximum of 20 subjects will be enrolled at up to 4 study centers. Subjects will attend a screening/pretreatment visit which may be performed on the same day as the treatment visit. Subjects may receive up to 5 treatments with the TempSure® Firm on the abdomen or flanks. All subjects will receive a phone call 1 week (1-10 days) post each treatment. Subjects may be asked to return for follow-up visits after their final treatment for incisional biopsies. A follow up may occur at 10, 20, and/or 30 days post their last treatment.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male or female between the age of 18 - 55 years old.
* Willing to receive treatments with the TempSure device and are willing to have biopsies taken from a control site and the treatment area.
* Understands and accepts obligation not to receive any other procedures on the treatment area through the length of the study.
* Understands and accepts the obligation and is logistically able to be present for all visits.
* Is willing to comply with all requirements of the study and sign the informed consent document.

Exclusion Criteria:

* Is pregnant or of childbearing potential and not using medically effective birth control, or has been pregnant in the last 3 months, currently breast feeding or planning a pregnancy during the study.
* The subject is currently enrolled in an investigational drug or device trial or has received an investigational drug or been treated with an investigational device within in the area to be treated 6 months prior to entering this study.
* The subject has a cut, wound, or infected skin on the area to be treated.
* The subject is on local, oral, or systemic anesthetic agents.
* The subject has any condition or is in a situation which in the investigators opinion may put the subject at significant risk, may confound study results or may interfere significantly with the subject's participation.
* The subject is currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within in the area to be treated 6 months (or at the discretion of the Investigator) prior to entering this study.

Cautionary Criteria:

* The subject has any embedded electronic device that gives or receives a signal, the device should be turned off or removed prior to treatment.
* The subject has an embedded pacemaker or implantable cardioverter defibrillator (ICD), the client's cardiologist must be consulted prior to treatment.

NOTE: This device has not been tested on patients implanted with electronic devices that receive or emit signals, such as: Pacemakers, Implantable Cardiac Defibrillators (ICD), or Cardiac Resynchronization Therapy (CRT) devices.

* If the neutral pad would need to be placed on a subject that has a metal plate, rod, or any metal implant that could conduct heat from the Smart Handpiece or surgical handpiece.
* The subject is allergic to adhesives, such as glues on medical tape, they should be alerted that a rash may occur on the neutral pad site and an over the counter solution may be used to treat the area.
* The subject is allergic to gold, such as the metallic covering of the TempSure handpieces.
* The subject is allergic to corn, such as the corn derivative ingredient in Parker Aquasonic Gel.
* If the subject has an unhealthy expectation of the results - this is not plastic surgery and all subject should be fully informed of the treatment's expected results.
* The subject has nerve insensitivity to heat in the treatment area.
* The subject has severe laxity or sagging that causes redundant folds of tissue or hanging skin in the area to be treated - this treatment will be ineffective.
* The subject has used Accutane (Isotretinoin) six to twelve months prior to treatment, as this can thin the skin and make it brittle.
* Studies of the use of the RF generator on subjects that have any of the following conditions is unknown:

  * Autoimmune Disease
  * Diabetic
  * Herpes Simplex
* Use caution when treating areas that have scars, tattoos, permanent makeup, and permanent brows.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Civiok, Study Director — Cynosure, Inc.
Locations (2):
- United States (2):
  - Bass Plastic Surgery PLLC, New York, New York
  - Aesthetic Pavilion, Staten Island, New York

IPD SHARING:
Plan to Share IPD: No
No data will be shared.

REFERENCES:
- [Background] Gupta V, Sharma VK. Skin typing: Fitzpatrick grading and others. Clin Dermatol. 2019 Sep-Oct;37(5):430-436. doi: 10.1016/j.clindermatol.2019.07.010. Epub 2019 Jul 17. PMID 31896400

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Biopsy Removed Post Tx
Started | 12
Completed | 0
Not Completed | 12

BASELINE CHARACTERISTICS:
Arm/Group | Biopsy Removed Post Tx
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants] — Population: 2 subjects did not have their ages analyzed.
  Participants
    number analyzed (Participants) | 10
    <=18 years | 0
    Between 18 and 65 years | 10
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One subject did not report their sex.
  Participants
    number analyzed (Participants) | 11
    Female | 11
    Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 5
  Middle Eastern | 1
  Caucasian | 5
  Asian | 1
FitzPatrick Skin Type [Count of Participants; unit: Participants] — Fitzpatrick Skin Types range from I-VI, with I representing the lowest amount of melanin (lightest skin) and VI representing the highest amount of melanin (darkest skin). Details on this scale can be found in the references section. Population: Only 5 subjects reported on their Fitzpatrick Skin Types.
  Participants
    number analyzed (Participants) | 5
    Fitzpatrick Skin Type I | 1
    Fitzpatrick Skin Type II | 0
    Fitzpatrick Skin Type III | 1
    Fitzpatrick Skin Type IV | 0
    Fitzpatrick Skin Type V | 1
    Fitzpatrick Skin Type VI | 2

OUTCOME MEASURES:

1. Primary Outcome: Histology of Biopsy
Description: Samples will be assessed independently and may be assessed for normal structures, cell viability, vascular injury, and overall morphologic traits, injury, and any indications of the healing response.
Time Frame: Up to 30 days post last treatment
Population: Data were not collected.
Arm/Group | Biopsy Removed Post Tx
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Subjects had their adverse event data collected from the beginning of the study, until the study was cancelled, an average of 1 month.
Arm/Group | Biopsy Removed Post Tx
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/99/NCT04584099/Prot_SAP_000.pdf